CLINICAL TRIAL: NCT01966536
Title: CD133+ Autologue Transplantation to Promote Ovarian Follicles Development in Women With Poor Ovarian Reserve.
Brief Title: CD133 Transplantation to Generate Oocytes in Poor Ovarian Reserve
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to fundamental changes in procedures design no patients have been enrolled
Sponsor: Hospital Universitario La Fe (Other)
Responsible Party: Principal Investigator, Dr. Antonio Pellicer Martínez, Doctor, Hospital Universitario La Fe
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Neofol2013
Record Dates: First submitted 2013-10-17; First posted 2013-10-21 (Estimated); Last update posted 2014-09-12 (Estimated); Status verified 2014-09

CONDITIONS: Ovarian Reserve

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Poor ovarian reserve (Experimental): Autologous transplantation of CD133+ cells into ovarian artery
  Interventions: Procedure: CD133+ cells transplantation into ovarian artery of one ovary

INTERVENTIONS:
Procedure: CD133+ cells transplantation into ovarian artery of one ovary

SUMMARY:
Women delay maternity and, as a consequence, available oocyte number and their quality decrease (9-18% of all IVF patients). Different treatment protocols have been developped nevertheless none of them optimal: the number of oocytes retrieved depends on the present ones. New generation of oocytes and follicles has been defended by some authors and bone marrow seems to be involved. What seems crucial is the niche that produces paracrine signals able to activate dormant cells and to attract undifferentiated cells from other tissues (homing). This phenomenon has been described by our group in other human reproductive tissues like endometrium. The purpose of the study is to improve ovarian reserve in unfertile women with poor ovarian reserve by means of bone marrow protective capacity.

CD133+ cells obtained from bone marrow will be delivered into the ovarian artery allowing them to colonize ovarian niche.

The study hypothesis is that CD133+ cells will improve ovarian reserve differentiating themselves into germ cells or, more likely, stimulating the niche to activate dormant follicles.

ELIGIBILITY:
Inclusion Criteria:

* < or= 40 years old
* FSH<15UI/L
* poor ovarian response after controlled ovarian stimulation with conventional doses (<3 oocytes) or two episodes of poor ovarian response after ovarian stimulation with maximal doses even if young or normal ovarian reserve study.
* Antral follicle count>2
* >1 antral follicle in the perfunded ovary
* AMH between 0,5 and 1pmol/L
* regular menstrual bleeding each 21-35 days
* To be candidate to autologous hematopoietic progenitors transplantation

Exclusion Criteria:

* Ovarian endometriosis
* Anovulation
* Any ovarian surgery considered risk factor of low ovarian response.
* Genetic factors associated to low ovarian response (Turner syndrome, FMR1 mutations...)
* Adquired conditions determining low response (chemotherapy, radiotherapy...)
* BMI > or = 30kg/m2
* Allergie to iodine
* Kidney failure

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2013-11; Primary Completion 2014-03 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Ovarian reserve | 6 months
  Measured by FSH-LH, oestradiol, AMH, antral follicle count

SECONDARY OUTCOMES:
Ovarian response to stimulation for oocyte retrieval | 6 months
  Number of MII oocytes obtained

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Pellicer, Doctor, Principal Investigator — Hospital Universitario La Fe
Locations (1):
- Hospital Universitario y Politécnico La Fe, Valencia, Valencia, Spain

REFERENCES:
- [Background] Munne S, Cohen J, Sable D. Preimplantation genetic diagnosis for advanced maternal age and other indications. Fertil Steril. 2002 Aug;78(2):234-6. doi: 10.1016/s0015-0282(02)03239-9. No abstract available. PMID 12137856
- [Background] Garcia-Velasco JA, Isaza V, Requena A, Martinez-Salazar FJ, Landazabal A, Remohi J, Pellicer A, Simon C. High doses of gonadotrophins combined with stop versus non-stop protocol of GnRH analogue administration in low responder IVF patients: a prospective, randomized, controlled trial. Hum Reprod. 2000 Nov;15(11):2292-6. doi: 10.1093/humrep/15.11.2292. PMID 11056121
- [Background] La Marca A, Sighinolfi G, Radi D, Argento C, Baraldi E, Artenisio AC, Stabile G, Volpe A. Anti-Mullerian hormone (AMH) as a predictive marker in assisted reproductive technology (ART). Hum Reprod Update. 2010 Mar-Apr;16(2):113-30. doi: 10.1093/humupd/dmp036. Epub 2009 Sep 30. PMID 19793843
- [Background] Johnson J, Canning J, Kaneko T, Pru JK, Tilly JL. Germline stem cells and follicular renewal in the postnatal mammalian ovary. Nature. 2004 Mar 11;428(6979):145-50. doi: 10.1038/nature02316. PMID 15014492
- [Background] White YA, Woods DC, Takai Y, Ishihara O, Seki H, Tilly JL. Oocyte formation by mitotically active germ cells purified from ovaries of reproductive-age women. Nat Med. 2012 Feb 26;18(3):413-21. doi: 10.1038/nm.2669. PMID 22366948
- [Background] Johnson J, Bagley J, Skaznik-Wikiel M, Lee HJ, Adams GB, Niikura Y, Tschudy KS, Tilly JC, Cortes ML, Forkert R, Spitzer T, Iacomini J, Scadden DT, Tilly JL. Oocyte generation in adult mammalian ovaries by putative germ cells in bone marrow and peripheral blood. Cell. 2005 Jul 29;122(2):303-15. doi: 10.1016/j.cell.2005.06.031. PMID 16051153
- [Background] Hong H, Yen HY, Brockmeyer A, Liu Y, Chodankar R, Pike MC, Stanczyk FZ, Maxson R, Dubeau L. Changes in the mouse estrus cycle in response to BRCA1 inactivation suggest a potential link between risk factors for familial and sporadic ovarian cancer. Cancer Res. 2010 Jan 1;70(1):221-8. doi: 10.1158/0008-5472.CAN-09-3232. Epub 2009 Dec 22. PMID 20028858
- [Background] Eggan K, Jurga S, Gosden R, Min IM, Wagers AJ. Ovulated oocytes in adult mice derive from non-circulating germ cells. Nature. 2006 Jun 29;441(7097):1109-14. doi: 10.1038/nature04929. Epub 2006 Jun 14. PMID 16799565
- [Background] Li J, Kawamura K, Cheng Y, Liu S, Klein C, Liu S, Duan EK, Hsueh AJ. Activation of dormant ovarian follicles to generate mature eggs. Proc Natl Acad Sci U S A. 2010 Jun 1;107(22):10280-4. doi: 10.1073/pnas.1001198107. Epub 2010 May 17. PMID 20479243
- [Background] Bhartiya D, Sriraman K, Parte S. Stem cell interaction with somatic niche may hold the key to fertility restoration in cancer patients. Obstet Gynecol Int. 2012;2012:921082. doi: 10.1155/2012/921082. Epub 2012 Apr 2. PMID 22548074
- [Background] Taylor HS. Endometrial cells derived from donor stem cells in bone marrow transplant recipients. JAMA. 2004 Jul 7;292(1):81-5. doi: 10.1001/jama.292.1.81. PMID 15238594
- [Background] Nagori CB, Panchal SY, Patel H. Endometrial regeneration using autologous adult stem cells followed by conception by in vitro fertilization in a patient of severe Asherman's syndrome. J Hum Reprod Sci. 2011 Jan;4(1):43-8. doi: 10.4103/0974-1208.82360. PMID 21772740
- [Background] Gargett CE, Healy DL. Generating receptive endometrium in Asherman's syndrome. J Hum Reprod Sci. 2011 Jan;4(1):49-52. PMID 21772741
- [Background] Zeng H, Li L, Chen JX. Overexpression of angiopoietin-1 increases CD133+/c-kit+ cells and reduces myocardial apoptosis in db/db mouse infarcted hearts. PLoS One. 2012;7(4):e35905. doi: 10.1371/journal.pone.0035905. Epub 2012 Apr 27. PMID 22558265
- [Background] Flesken-Nikitin A, Hwang CI, Cheng CY, Michurina TV, Enikolopov G, Nikitin AY. Ovarian surface epithelium at the junction area contains a cancer-prone stem cell niche. Nature. 2013 Mar 14;495(7440):241-5. doi: 10.1038/nature11979. Epub 2013 Mar 6. PMID 23467088